CLINICAL TRIAL: NCT05341011
Title: Establishment of Social Skills Training Group in Adolescents With Autism Spectrum Disorder and Effectiveness Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201906022RIND
Record Dates: First submitted 2022-03-31; First posted 2022-04-22 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder High-Functioning
Keywords: autism spectrum disorder; social skills training program; adolescents
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (TX) Group (Experimental): The TX group received 14 weeks of the PEERS® intervention immediately following a baseline assessment,
  Interventions: Behavioral: PEERS® Social Skills Training
- Delayed Treatment Control (DTC) Group (Experimental): The DTC group received the same intervention after a 14-week waiting period. Parents and teens attended concurrent sessions held in separate rooms.
  Interventions: Behavioral: PEERS® Social Skills Training

INTERVENTIONS:
Behavioral: PEERS® Social Skills Training — The PEERS® consisted of 14 weekly 90-min didactic sessions. Adolescents and their parents attended separate concurrent sessions.
  Each session began with a review of the homework assignment from the previous week and allowed time for troubleshooting problems encountered in completing the behavioral assignment. This was followed by a didactic lesson on the weekly topic. Didactic lessons included content related to various social skills and peer interactions. Parents attendance was a mandatory component of PEERS® intervention. Parents were expected to enhance generalization of social skills through in vivo social coaching in natural social settings and increase homework compliance as well as practice of newly learned social skills. A 10-min reunification between adolescents and caregivers was arranged at the end of each session to review the skills taught in the session and assign corresponding homework for the next session.

SUMMARY:
Autism spectrum disorders (ASD) is a neurodevelopmental disorder characterized by persistent deficits in social communication and social interaction, and the presence of restricted, repetitive behavior and interests. Their social relationships with peers may remain a challenge or even worsen for individuals with ASD throughout the school years and beyond. Adolescence may be a particularly difficult developmental period, as they may have greater motivation or desire to engage with peers but also have greater awareness of their social disability. Adolescents with ASD are reported to experience greater loneliness and mood disturbances, and have poorer friendship quality and social network status than their typically developing peers. Moreover, a growing body of literature indicating that students with ASD have increased risk at all kinds of bullying involvement. These findings underscore the importance of providing social skills training. One of the empirically supported intervention program that targets adolescents with ASD is the Program for the Education and Enrichment of Relational Skills (PEERS®). This is a parent-assisted, manualized social skills training program that addresses crucial areas of social functioning for adolescents. Psycho-education and cognitive-behavioral therapy techniques are employed to help adolescents develop ecologically valid skills for making and maintaining friendships. Moreover, caregiver attendance at the same time in the caregiver group was a mandatory component to enhance the child/s generalization of social skills.

Adolescents with ASD and normal IQ will be recruit to attend the 14-week PEERS® group training together with a parent. The participants will be stratified by gender and randomized to a treatment (TX) group or delayed treatment control (DTC) group. A team member uninvolved in the program made the random allocation with random digit generated by computer.

This study investigated the acceptability, feasibility and effectiveness of the Taiwanese adolescent PEERS® program.

DETAILED DESCRIPTION:
The PEERS® group will be run by PI and the special education teacher (one is the leader for teen session and the other is the leader for parent session) both with substantial experience conducting social skills programs for children and adolescents, and parent education groups related to ASD, under the on-site supervision of co-PI with comprehensive training through the UCLA PEERS® Clinic by the program developer. Three research assistants (one is a psychiatrist, another is an occupational therapist, and the other is a social worker) will take the part of role-play (following the social scenario script) during PEERS® intervention.

The TX group received 14 weeks of the PEERS® intervention immediately following a baseline assessment, while the DTC group received the same intervention after a 14-week waiting period. Parents and teens attended concurrent sessions held in separate rooms.

ELIGIBILITY:
Inclusion Criteria:

* Teens:

  1. currently enrolled in school
  2. clinical diagnosis of Autism Spectrum Disorder (ASD)
  3. experiencing social difficulties
  4. scored ≧ 26 on the caregiver-reported Autism Spectrum Quotient (AQ)
  5. verbal fluency in Chinese
  6. with a full-scale IQ > 70 on WAIS-IV
  7. with motivation to participate in the intervention
* Parents:

  1. verbal fluency in Chinese
  2. with motivation to participate in the intervention

Exclusion Criteria:

1. major mental illness
2. sever visual or hearing impairment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Test of Adolescents Social Skills Knowledge (TASSK) | Baseline and Pre-Intervention
  The TASSK consists of 26 items derived from the 13 didactic lessons in PEERS® to assess the specific social skills knowledge taught during the intervention. Adolescents were asked to read sentence stems and choose the best answer from two options to complete the sentence in each item. Each correct answer was awarded one point. Higher scores on this task reflected better knowledge of social etiquette, and the maximum possible score was 26. Previous studies on the PEERS® intervention have shown that the TASSK is sensitive to treatment effects. The original English Version was reported a coefficient alpha of 0.56, and the Chinese version (Shum et al., 2019) also obtained a ronbach's alpha of 0.50. The reliability of this measure was thus similar to those reported in previous studies.
Test of Adolescents Social Skills Knowledge (TASSK) | During the Intervention
  The TASSK consists of 26 items derived from the 13 didactic lessons in PEERS® to assess the specific social skills knowledge taught during the intervention. Adolescents were asked to read sentence stems and choose the best answer from two options to complete the sentence in each item. Each correct answer was awarded one point. Higher scores on this task reflected better knowledge of social etiquette, and the maximum possible score was 26. Previous studies on the PEERS® intervention have shown that the TASSK is sensitive to treatment effects. The original English Version was reported a coefficient alpha of 0.56, and the Chinese version (Shum et al., 2019) also obtained a ronbach's alpha of 0.50. The reliability of this measure was thus similar to those reported in previous studies.
Test of Adolescents Social Skills Knowledge (TASSK) | Immediately after the Intervention
  The TASSK consists of 26 items derived from the 13 didactic lessons in PEERS® to assess the specific social skills knowledge taught during the intervention. Adolescents were asked to read sentence stems and choose the best answer from two options to complete the sentence in each item. Each correct answer was awarded one point. Higher scores on this task reflected better knowledge of social etiquette, and the maximum possible score was 26. Previous studies on the PEERS® intervention have shown that the TASSK is sensitive to treatment effects. The original English Version was reported a coefficient alpha of 0.56, and the Chinese version (Shum et al., 2019) also obtained a ronbach's alpha of 0.50. The reliability of this measure was thus similar to those reported in previous studies.
Test of Adolescents Social Skills Knowledge (TASSK) | Change from Post-Intervention at 4 months
  The TASSK consists of 26 items derived from the 13 didactic lessons in PEERS® to assess the specific social skills knowledge taught during the intervention. Adolescents were asked to read sentence stems and choose the best answer from two options to complete the sentence in each item. Each correct answer was awarded one point. Higher scores on this task reflected better knowledge of social etiquette, and the maximum possible score was 26. Previous studies on the PEERS® intervention have shown that the TASSK is sensitive to treatment effects. The original English Version was reported a coefficient alpha of 0.56, and the Chinese version (Shum et al., 2019) also obtained a ronbach's alpha of 0.50. The reliability of this measure was thus similar to those reported in previous studies.
Test of Adolescents Social Skills Knowledge (TASSK) | Change from Post-Intervention at 8 months
  The TASSK consists of 26 items derived from the 13 didactic lessons in PEERS® to assess the specific social skills knowledge taught during the intervention. Adolescents were asked to read sentence stems and choose the best answer from two options to complete the sentence in each item. Each correct answer was awarded one point. Higher scores on this task reflected better knowledge of social etiquette, and the maximum possible score was 26. Previous studies on the PEERS® intervention have shown that the TASSK is sensitive to treatment effects. The original English Version was reported a coefficient alpha of 0.56, and the Chinese version (Shum et al., 2019) also obtained a ronbach's alpha of 0.50. The reliability of this measure was thus similar to those reported in previous studies.
Test of Adolescents Social Skills Knowledge (TASSK) | Change from Post-Intervention at 16 months
  The TASSK consists of 26 items derived from the 13 didactic lessons in PEERS® to assess the specific social skills knowledge taught during the intervention. Adolescents were asked to read sentence stems and choose the best answer from two options to complete the sentence in each item. Each correct answer was awarded one point. Higher scores on this task reflected better knowledge of social etiquette, and the maximum possible score was 26. Previous studies on the PEERS® intervention have shown that the TASSK is sensitive to treatment effects. The original English Version was reported a coefficient alpha of 0.56, and the Chinese version (Shum et al., 2019) also obtained a ronbach's alpha of 0.50. The reliability of this measure was thus similar to those reported in previous studies.
Quality of Play Questionnaire (QPQ) | Baseline and Pre-Intervention
  The QPQ was adapted from Frankel and Mintz (2011) and included in the original treatment manual as QPQ-P (parent) and QPQ-A (adolescent). Parents and adolescents were asked to complete the questionnaire independently. There are 12 items in the questionnaire, 2 of which assess the frequency of get-togethers over the previous month, and the remaining 10 items gauge the level of conflict during the last hosted get-together. Items on the Conflict Scale, for instance, include "They/We criticized or teased each other". Higher scores on the Conflict Scale indicated more conflict observed during the last get-together.
Quality of Play Questionnaire (QPQ) | During the Intervention
  The QPQ was adapted from Frankel and Mintz (2011) and included in the original treatment manual as QPQ-P (parent) and QPQ-A (adolescent). Parents and adolescents were asked to complete the questionnaire independently. There are 12 items in the questionnaire, 2 of which assess the frequency of get-togethers over the previous month, and the remaining 10 items gauge the level of conflict during the last hosted get-together. Items on the Conflict Scale, for instance, include "They/We criticized or teased each other". Higher scores on the Conflict Scale indicated more conflict observed during the last get-together.
Quality of Play Questionnaire (QPQ) | Immediately after the Intervention
  The QPQ was adapted from Frankel and Mintz (2011) and included in the original treatment manual as QPQ-P (parent) and QPQ-A (adolescent). Parents and adolescents were asked to complete the questionnaire independently. There are 12 items in the questionnaire, 2 of which assess the frequency of get-togethers over the previous month, and the remaining 10 items gauge the level of conflict during the last hosted get-together. Items on the Conflict Scale, for instance, include "They/We criticized or teased each other". Higher scores on the Conflict Scale indicated more conflict observed during the last get-together.
Quality of Play Questionnaire (QPQ) | Change from Post-Intervention at 4 months
  The QPQ was adapted from Frankel and Mintz (2011) and included in the original treatment manual as QPQ-P (parent) and QPQ-A (adolescent). Parents and adolescents were asked to complete the questionnaire independently. There are 12 items in the questionnaire, 2 of which assess the frequency of get-togethers over the previous month, and the remaining 10 items gauge the level of conflict during the last hosted get-together. Items on the Conflict Scale, for instance, include "They/We criticized or teased each other". Higher scores on the Conflict Scale indicated more conflict observed during the last get-together.
Quality of Play Questionnaire (QPQ) | Change from Post-Intervention at 8 months
  The QPQ was adapted from Frankel and Mintz (2011) and included in the original treatment manual as QPQ-P (parent) and QPQ-A (adolescent). Parents and adolescents were asked to complete the questionnaire independently. There are 12 items in the questionnaire, 2 of which assess the frequency of get-togethers over the previous month, and the remaining 10 items gauge the level of conflict during the last hosted get-together. Items on the Conflict Scale, for instance, include "They/We criticized or teased each other". Higher scores on the Conflict Scale indicated more conflict observed during the last get-together.
Quality of Play Questionnaire (QPQ) | Change from Post-Intervention at 16 months
  The QPQ was adapted from Frankel and Mintz (2011) and included in the original treatment manual as QPQ-P (parent) and QPQ-A (adolescent). Parents and adolescents were asked to complete the questionnaire independently. There are 12 items in the questionnaire, 2 of which assess the frequency of get-togethers over the previous month, and the remaining 10 items gauge the level of conflict during the last hosted get-together. Items on the Conflict Scale, for instance, include "They/We criticized or teased each other". Higher scores on the Conflict Scale indicated more conflict observed during the last get-together.
Chinese version of the School Bullying Experience Questionnaire (C-SBEQ) | Baseline and Pre-Intervention
  The self-reported C-SBEQ was used to evaluate participants' involvement in school bullying in recent months with 16 items answered on a Likert 4-point scale range with 0 indicating "never", 1 indicating "just a little", 2 indicating "often", and 3 indicating "all the time". This scale was composed of four 4-item subscales evaluating being a victim of passive bullying (items 1 to 4, including social exclusion, being called a mean nickname, and being spoken ill of), being a victim of active bullying (items 5 to 8, including being beaten up, being forced to do work, and having money, school supplies, and snacks taken away), being a perpetrator of passive bullying (items 9 to 12), and being a perpetrator of active bullying (items 13 to 16).
Chinese version of the School Bullying Experience Questionnaire (C-SBEQ) | During the Intervention
  The self-reported C-SBEQ was used to evaluate participants' involvement in school bullying in recent months with 16 items answered on a Likert 4-point scale range with 0 indicating "never", 1 indicating "just a little", 2 indicating "often", and 3 indicating "all the time". This scale was composed of four 4-item subscales evaluating being a victim of passive bullying (items 1 to 4, including social exclusion, being called a mean nickname, and being spoken ill of), being a victim of active bullying (items 5 to 8, including being beaten up, being forced to do work, and having money, school supplies, and snacks taken away), being a perpetrator of passive bullying (items 9 to 12), and being a perpetrator of active bullying (items 13 to 16).
Chinese version of the School Bullying Experience Questionnaire (C-SBEQ) | Immediately after the Intervention
  The self-reported C-SBEQ was used to evaluate participants' involvement in school bullying in recent months with 16 items answered on a Likert 4-point scale range with 0 indicating "never", 1 indicating "just a little", 2 indicating "often", and 3 indicating "all the time". This scale was composed of four 4-item subscales evaluating being a victim of passive bullying (items 1 to 4, including social exclusion, being called a mean nickname, and being spoken ill of), being a victim of active bullying (items 5 to 8, including being beaten up, being forced to do work, and having money, school supplies, and snacks taken away), being a perpetrator of passive bullying (items 9 to 12), and being a perpetrator of active bullying (items 13 to 16).
Chinese version of the School Bullying Experience Questionnaire (C-SBEQ) | Change from Post-Intervention at 4 months
  The self-reported C-SBEQ was used to evaluate participants' involvement in school bullying in recent months with 16 items answered on a Likert 4-point scale range with 0 indicating "never", 1 indicating "just a little", 2 indicating "often", and 3 indicating "all the time". This scale was composed of four 4-item subscales evaluating being a victim of passive bullying (items 1 to 4, including social exclusion, being called a mean nickname, and being spoken ill of), being a victim of active bullying (items 5 to 8, including being beaten up, being forced to do work, and having money, school supplies, and snacks taken away), being a perpetrator of passive bullying (items 9 to 12), and being a perpetrator of active bullying (items 13 to 16).
Chinese version of the School Bullying Experience Questionnaire (C-SBEQ) | Change from Post-Intervention at 8 months
  The self-reported C-SBEQ was used to evaluate participants' involvement in school bullying in recent months with 16 items answered on a Likert 4-point scale range with 0 indicating "never", 1 indicating "just a little", 2 indicating "often", and 3 indicating "all the time". This scale was composed of four 4-item subscales evaluating being a victim of passive bullying (items 1 to 4, including social exclusion, being called a mean nickname, and being spoken ill of), being a victim of active bullying (items 5 to 8, including being beaten up, being forced to do work, and having money, school supplies, and snacks taken away), being a perpetrator of passive bullying (items 9 to 12), and being a perpetrator of active bullying (items 13 to 16).
Chinese version of the School Bullying Experience Questionnaire (C-SBEQ) | Change from Post-Intervention at 16 months
  The self-reported C-SBEQ was used to evaluate participants' involvement in school bullying in recent months with 16 items answered on a Likert 4-point scale range with 0 indicating "never", 1 indicating "just a little", 2 indicating "often", and 3 indicating "all the time". This scale was composed of four 4-item subscales evaluating being a victim of passive bullying (items 1 to 4, including social exclusion, being called a mean nickname, and being spoken ill of), being a victim of active bullying (items 5 to 8, including being beaten up, being forced to do work, and having money, school supplies, and snacks taken away), being a perpetrator of passive bullying (items 9 to 12), and being a perpetrator of active bullying (items 13 to 16).

SECONDARY OUTCOMES:
Swanson, Nolan, and Pelham, version IV (SNAP-IV) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Chinese version of the SNAP-IV is a 26-item scale using a 4-point Likert scale with a score of 0 for "not at all," 1 for "just a little," 2 for "quite a bit," and 3 for "very much." It contains 18 items according to the core symptoms based on the ADHD and ODD criteria in the DSM-IV. The norm and psychometric properties of the Chinese SNAP-IV have been established (Gau et al., 2008), and have been extensively used to assess ADHD and ODD symptoms in clinical and research settings. It has been widely used in many studies in Taiwan. We used symptom-count criterion from the full diagnostic criteria stated in the DSM-IV. A score of 2 (quite a bit) or 3 (very much) in each item was coded as the symptomatic presence of this behavior and 0 (not at all) or 1 (just a little) as absence in this study.
Social Adjustment Inventory for Children and Adolescents (SAICA) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Social Adjustment Inventory for Children and Adolescents (SAICA) is a semi-structured interview designed to assess the adaptive functioning of youths aged 6-18 in 4 major role areas, including school, spare time activities, peer relations, and home behaviors reported by the youths themselves or by their parents. The youths with higher score had either poorer functioning or more severe problems in the assessed domain. The Chinese version of the SAICA has good psychometric properties and is widely used in assessing social functions in Taiwan.
Empathy Quotient (EQ) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Empathy Quotient (EQ) is a parent-report measure of empathy. Around 81% of adolescents with ASD score less than 30 on the EQ, compared to 12% of controls; the groups together report excellent internal consistency (.92) and test-retest reliability (.97). The Chinese version of EQ has satisfactory reliability and validity (Huang HY, Gau SS, unpublished). The EQ will be administered to caregivers at baseline, post-treatment to assess treatment outcome.
Friendship Questionnaire (FQ) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Friendship Questionnaire (FQ) is a self-report questionnaire comprises 35 questions, on 27 of which it is possible to score. Questions were taken from the sex differences literature above. Although this may sound circular, the aim of this study was to investigate whether a quantitative self-report questionnaire would produce the same results as previous observational studies. The maximum score for each item on the FQ is 5 points, with fewer points also available for some items. The Chinese version of FQ has satisfactory reliability and validity.
Friendship Quality Scale (FQS) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Friendship Qualities Scale is a theoretically grounded, multidimensional measurement instrument to assess the quality of children's and early adolescents' relationships with their best friends according to 5 conceptually meaningful aspects of the friendship relation. These dimensions are companionship, conflict, help/aid, security and closeness. FQS's items are commonly statements about how meaningful adolescents with their friends in five points Likert scale, ranged from 1 (definitely not true) to 5 (definitely true) with the items are mentioned like, "if I have a problem at school or at home I can talk to my friend about it." FQS's score is obtained through the calculation of each participant's average from 32 items Scores on items within each dimension are averaged to yield composite scores measuring each dimension. A total score was computed as the average of the five domain scores (conflict score reversed).
Assessing Emotions Scale (AES) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Assessing Emotions Scale (AES), also named as the Schutte Emotional Intelligence Scale, is a 33-item self-report inventory focusing on typical emotional intelligence. This scale, based on Salovey and Mayer's (1990) original model of emotional intelligence that proposes emotional intelligence consists of appraisal of emotion in the self and others, expression of emotion, regulation of emotion in the self and others, and utilization of emotion in solving problems, attempts to assess characteristic, or trait, emotional intelligence. Respondents rate themselves on the items using a 5-point scale. Respondents require on average five minutes to complete the scale.
Youth Self Report (YSR) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Youth Self Report (YSR) is a 112-item self-report designed for children and adolescents aged 11-18, that assesses behavioral competency and behavioral problems. The Chinese versions of the YSR used in Taiwan was based on the 1991 versions. A total of 83 items were retained to create eight narrow-band behavioral/emotional problem syndromes for the YSR, including attention problems, anxious/depressed symptoms, aggressive behaviors, delinquent behaviors, social problems, somatic complaints, thought problems, and withdraw. The reliability and validity of the Chinese versions of the YSR has been demonstrated previously in Taiwan, and the scale has been widely used to measure emotional and behavioral problems in Taiwanese research. The standard scores are scaled so that 50 is average for the youth's age and gender, with a standard deviation of 10 points. Higher scores indicate greater problems.
Child Behavior Checklist (CBCL) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Child Behavior Checklist (CBCL) which is a standardized parent-report questionnaire rating scale assessing a broad range of psychopathology in children aged 4-18. The Chinese versions of the CBCL used in Taiwan was based on the 1991 versions. A total of 83 items were retained to create eight narrow-band behavioral/emotional problem syndromes for the CBCL, including attention problems, anxious/depressed symptoms, aggressive behaviors, delinquent behaviors, social problems, somatic complaints, thought problems, and withdraw. The reliability and validity of the Chinese versions of the CBCL have been demonstrated previously in Taiwan, and the scale has been widely used to measure emotional and behavioral problems in Taiwanese research. The standard scores are scaled so that 50 is average for the youth's age and gender, with a standard deviation of 10 points. Higher scores indicate greater problems.
World Health Organization Quality of Life (WHOQoL-BREF) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The brief version of the World Health Organization's Quality of Life (WHOQOL-BREF) contains two items from the Overall Quality of Life and General Health facet and one item from each of the remaining 24 facets. These facets are categorized into four major domains: Physical Capacity (7 items), Psychological Well-being (6 items), Social Relationships (3 items), and Environment (8 items). The Taiwanese version of the WHOQOL-BREF was developed in compliance with WHO guidelines with satisfactory reliability and validity. In addition to comprising 26 items translated from the original WHOQOL-BREF, the Taiwanese version includes two additional items of local importance, i.e. being respected and food availability. The two local items are categorized into the Social relationships (being respected) and Environment (food availability) domains, respectively.
Parenting Stress Index - Short Form (PSI-SF) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Parenting Stress Index - Short Form (PSI-SF) was used to assess parenting stress. All 36 items on the PSI-SF was written at a 5-point Likert-type scale with 1 indicating (strongly disagree) and 5 indicating (strongly agree). Child and parent domains combine to form total stress scale. The Chinese version has good psychometric properties and has been commercialized. The PSI-SF yields a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The Chinese version has good psychometric properties and has been commercialized.
Parental Bonding Instrument (PBI) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Parental Bonding Instrument (PBI) is a 25-item instrument that measures parenting styles during the child's first 16 years, with three principal dimensions: care/affection (12 items), overprotection (7 items) and authoritarianism (6 items) . A high score on the care/affection subscale reflects affection and warmth. Overprotection reflects overprotective parenting and denial of the child's psychological autonomy, and authoritarianism reflects parental authoritarian control over the child's behavior. The psychometric properties of the Chinese PBI have been described elsewhere.
Communicative Behavior Observatory Scale (CBOS) Behavior Observatory Scale (CBOS) | During the Intervention
  The Communicative Behavior Observatory Scale (CBOS) is a 10-item observer-rated scale designed to assess communicative behaviors during interpersonal interaction for individuals with ASD. Observers rated the items on a nine-point scale according to the frequency of the behaviors. Items include: (1) keeps appropriate distance during conversation, (2) keeps eye contact during conversation, (3) appropriate nodding/shaking head/gestures, (4) maintains conversation appropriately, (5) switches conversation topics appropriately, (6) appropriate amount of voice/intonation, (7) appropriate facial expression when talking, (8) reciprocity during conversation, (9) emotional regulation, and (10) overall communicative behaviors.
Social Responsiveness Scale (SRS) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Social Responsiveness Scale (SRS) is a 65-item rating scale of the severity of ASD symptoms as they occur in natural settings. It provides a clinical representation of an individual's social impairments, assessing social awareness, social information processing, capacity for reciprocal social communication, social avoidance, and autistic mannerisms using T-scores (M = 50; SD =10). Higher scores on the SRS reflect greater impairment and autistic symptoms with scores >= 60 in the clinical threshold. The Chinese-language SRS has demonstrated a satisfactory four-factor structure with high internal consistency (Cronbach's alpha, .94-.95), i.e., social communication, autistic mannerism, social awareness, and social emotion. The Chinese SRS has been widely used to assess autistic traits in Taiwan.
Autism Spectrum Quotient (AQ) | Baseline and Pre-Intervention, immediate Post-Intervention, and the 4th-, 8th- and 16th-month follow-up
  The Autism Spectrum Quotient (AQ) (Baron-Cohen, Wheelwright, Skinner, Martin, & Clubley, 2001) is a 50-item scale that measures autistic traits along five subscales: social skills, attention shifting, attention to detail, communication, and imagination. There are 3 versions of AQ, which is AQ-child, AQ-Adolescent, and AQ-Adult. The AQ-Child is a parent-report questionnaire developed to detect autistic traits in children at 4-11 years of age, and the AQ-Adolescent is also a parent-report questionnaire for age at 12-15 years, and the AQ-Adult is the self- and parent-report scale for aged 16 years old and above. Each item of the questionnaire is rated on a four-point scale with answer categories of "almost always true", "often true", "sometimes true" and "not true". The AQ in Chinese-language has been used to measure autistic traits in Taiwan.
Autism Diagnostic Observation Schedule (ADOS) | Baseline and Pre-Intervention and immediate Post-Intervention
  The Autism Diagnostic Observation Schedule (ADOS) is a standard instrument for diagnosing and assessing autism, consists of a series of structured and semi-structured tasks that involve social interaction between the examiner and the subject. Through the tasks, the examiner observes and rates the subject's social and communication behaviors relevant to the diagnosis of autism. Four modules are developed for subjects with different age and verbal ability, here we will apply Module 4 for adolescent with fluent speech. The ADOS algorithm has been translated into Chinese by a group of child psychiatrists lead by Co-PI Gau SS.
Autism Diagnostic Interview-Revised (ADI-R) | Baseline
  The Autism Diagnostic Interview-Revised (ADI-R) is a standardized, comprehensive, semi-structured, investigator-based interview of the caregivers. It covers most developmental and behavioral aspects of ASD, including reciprocally social interaction, communication, and repetitive behaviors and stereotyped patterns, for children with a mental age from about 18 months into adulthood. The Chinese version of the ADI-R was approved by the World Psychological Association in 2007 and has been extensively used in ASD research in Taiwan.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Ni Hsiao, MA, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Some participants clearly stated that they don't want their data to be shared.

REFERENCES:
- [Background] Laugeson EA, Frankel F, Gantman A, Dillon AR, Mogil C. Evidence-based social skills training for adolescents with autism spectrum disorders: the UCLA PEERS program. J Autism Dev Disord. 2012 Jun;42(6):1025-36. doi: 10.1007/s10803-011-1339-1. PMID 21858588
- [Background] Laugeson EA, Frankel F, Mogil C, Dillon AR. Parent-assisted social skills training to improve friendships in teens with autism spectrum disorders. J Autism Dev Disord. 2009 Apr;39(4):596-606. doi: 10.1007/s10803-008-0664-5. Epub 2008 Nov 18. PMID 19015968
- [Background] Rao PA, Beidel DC, Murray MJ. Social skills interventions for children with Asperger's syndrome or high-functioning autism: a review and recommendations. J Autism Dev Disord. 2008 Feb;38(2):353-61. doi: 10.1007/s10803-007-0402-4. Epub 2007 Jul 20. PMID 17641962
- [Background] Schroeder JH, Cappadocia MC, Bebko JM, Pepler DJ, Weiss JA. Shedding light on a pervasive problem: a review of research on bullying experiences among children with autism spectrum disorders. J Autism Dev Disord. 2014 Jul;44(7):1520-34. doi: 10.1007/s10803-013-2011-8. PMID 24464616
- [Background] Andanson J, Pourre F, Maffre T, Raynaud JP. [Social skills training groups for children and adolescents with Asperger syndrome: A review]. Arch Pediatr. 2011 May;18(5):589-96. doi: 10.1016/j.arcped.2011.02.019. Epub 2011 Apr 1. French. PMID 21458972
- [Background] Yoo HJ, Bahn G, Cho IH, Kim EK, Kim JH, Min JW, Lee WH, Seo JS, Jun SS, Bong G, Cho S, Shin MS, Kim BN, Kim JW, Park S, Laugeson EA. A randomized controlled trial of the Korean version of the PEERS((R)) parent-assisted social skills training program for teens with ASD. Autism Res. 2014 Feb;7(1):145-61. doi: 10.1002/aur.1354. Epub 2014 Jan 9. PMID 24408892
- [Derived] Hsiao MN, Chien YL, Tai YM, Chen HM, Shih HH, Chen LW, Chen YY, Soong WT, Chiu YN, Tsai WC, Laugeson E, Tseng MH, Gau SS. A preliminary randomized controlled study of the PEERS(R) program for Taiwanese autistic adolescents: The effectiveness on reducing school bullying and enhancing social function. Autism Res. 2024 Aug;17(8):1705-1720. doi: 10.1002/aur.3213. PMID 39169699